CLINICAL TRIAL: NCT06241092
Title: AI-Based Multimodal Multi-tasks Analysis Reveals Tumor Molecular Heterogeneity, Predicts Preoperative Lymph Node Metastasis and Prognosis in Papillary Thyroid Carcinoma: A Retrospective Study
Brief Title: AI-Based Multimodal Multi-tasks Analysis Reveals Tumor Molecular Heterogeneity, Predicts Preoperative Lymph Node Metastasis and Prognosis in Papillary Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yunfang Yu, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2021-259
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Papillary Thyroid Carcinoma; Molecular Heterogeneity; Multi-model Analysis; Artificial Intelligence; Lymph Node Metastases; Disease-free Survival
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCGA
- SYSMH

INTERVENTIONS:
Other:

SUMMARY:
This study involved a comprehensive analysis of 256 PTC patients from Sun Yat-sen Memorial Hospital of Sun Yat-sen University (SYSMH) and 499 patients from The Cancer Genome Atlas. DNA-based next-generation sequencing (NGS) and single-cell RNA sequencing (scRNA-seq) were employed to capture genetic alterations and TME heterogeneity. A deep learning multimodal model was developed by incorporating matched histopathology slide images, genomic, transcriptomic, immune cells data to predict LNM and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age Diagnosis of Papillary thyroid carcinoma at least one months before trial Willing to return for required follow-up (posttest) visits

Exclusion Criteria:

The patient requires valve or other likely surgery The patient is unable to carry out any physical activity without discomfort The patient had thyroid ache within three months prior to enrollment The patient refuses to give informed consent The patient is a candidate for coronary bypass surgery or something similar

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis | 2021.10.1
  Lymph node metastasis is frequently influenced by a myriad of factors, and tumor heterogeneity stands out as a significant contributing element.

SECONDARY OUTCOMES:
Disease-free survival | 2021.10.1
  Disease-free survival is defined as the time from randomization to the first occurrence of a relapse, progression, or death from any cause, commonly used in clinical trials of adjuvant therapy after curative surgery or radiation therapy. It is also used as a primary endpoint in studies of neoadjuvant therapy and a useful endpoint for evaluating the efficacy of treatments that aim to prevent cancer recurrence research

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China